CLINICAL TRIAL: NCT00546468
Title: Prospective Randomized Trial of Laparoscopy-assisted Distal Gastrectomy (LADG) Versus Open Distal Gastrectomy (ODG) in Patients With Early Gastric Cancer (EGC)
Brief Title: Clinical Study on Laparoscopic Gastrectomy for Early Gastric Cancer (COACT_0301)
Acronym: NCC052
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Woo Kim, Head of Department of Gastric Cancer Surgery, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: _NCCCTS-052
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Gastric Cancer
Keywords: stomach cancer; laparoscopy; gastrectomy; QOL; survival; clinical study
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopy assisted distal gastrectomy (Experimental): Laparoscopy assisted distal gastrectomy with D2 lymph node dissection.Surgery will be done in similar operative extent with control open distal gastrectomy. Omentectomy will be omitted.
  Interventions: Procedure: laparoscopy assisted distal gastrectomy
- Open Distal Gastrectomy (Active Comparator): Conventional standard D2 open distal gastrectomy without omentectomy.
  Interventions: Procedure: Open distal gastrectomy

INTERVENTIONS:
Procedure: laparoscopy assisted distal gastrectomy — under general endotracheal anesthesia, Five laparoscopic ports are made. Lymph node dissection and ligations of vessels are done in laparoscopic field. A 5-6cm small incision is made transversely in RUQ of the abdomen. Through the incisional window, stomach is taken out and resected. A Billroth I gastroduodenostomy using EEA stapler and GIA is performed. Abdomen is closed after hemostasis.
  Other Names: LADG
  Arms: Laparoscopy assisted distal gastrectomy
Procedure: Open distal gastrectomy — Open distal gastrectomy is performed under general endotracheal anesthesia. A long midline incision is made. omentectomy is skipped and D2 lymph node dissection is performed. Anastomosis is done in same manner as LADG. Abdomen is closed after hemostasis
  Other Names: ODG
  Arms: Open Distal Gastrectomy

SUMMARY:
Rationale: For the treatment of early gastric cancer (EGC) in the distal portion of the stomach, subtotal gastrectomy and lymph node dissection has been a standard operation. With the increasing tendency toward minimally invasive surgery, there has been an effort to apply minimally invasive techniques to the treatment of EGC. Laparoendoluminal mucosectomy and lesion-lifting gastric wedge resection have been developed for this purpose. However, these methods have the disadvantage of limited indications according to the size, shape and depth of invasion. Kitano et al. performed the first laparoscopy-assisted subtotal gastrectomy with lymph node dissection and manual anastomosis with anterior wall lifting method for a patient with EGC. In 1995, Uyama et al. and Nagai et al. performed laparoscopy-assisted subtotal gastrectomy with lymph node dissections using an automatic stapler instead of manual anastomosis for the gastroduodenal anastomosis. It has been possible to maintain an adequate distance from the lesion to the proximal and distal margins of resection, to perform radical lymph node dissection, and to achieve excellent postoperative recovery. However, there is a very limited evidence of superiority of laparoscopic gastrectomy over open surgery. There is only one interim report of randomized clinical trial of comparing laparoscopic gastrectomy and open gastrectomy. A well-designed clinical study to prove the benefit and safety is definitely needed Objective: to compare Laparoscopy - assisted Distal Gastrectomy (LADG) with Open Distal Gastrectomy (ODG) in terms of survival, recovery, pain, complications, and quality of life (QOL) Hypothesis: LADG is beneficial in QOL, pain, recovery, complications while maintaining equivalent survival with ODG

DETAILED DESCRIPTION:
1. Randomization

   Randomization is done by person who is not involved in study. So it is done by the person in Center for Clinical Trial in National Cancer Center. The patient is enrolled in the out-patient clinic after getting informed consent of the clinical study from the patient. Surgeon factor is not considered as a randomization factor because this clinical study will be performed intramurally. In Center for Gastric Cancer, National Cancer Center, Surgical techniques and extent of resections are generally standardized and surgical outcomes are same in terms of complication and recovery.
2. Follow-up schedule

   Patients are followed up in the outpatient department at four weeks, three months, six months, and twelve months after the operation, and every six months thereafter. On each visit, history was reviewed and physical examination was done. A complete blood count (CBC) and serum chemistry were evaluated also. An esophago-gastro-duodenoscopy (EGD) was performed at three months after the operation and yearly thereafter. Abdominal computed tomography (ACT) was evaluated annually.
3. Assessment of QOL The European EORTC QLQ-C30 (version 3.0) questionnaire is a 30-item cancer-specific integrated system for assessing the health-related QOL of cancer patients. The questionnaire incorporates five scales of function (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea and vomiting), a global health and QOL scale, and single items for the assessment of additional symptoms commonly reported by cancer patients (e.g., dyspnea, appetite loss, sleep disturbance, constipation and diarrhea), as well as the perceived financial impact of the disease and treatment. All items were scored on four-point Likert scales, with the exception of two items in the global health QOL scale, which used modified seven-point linear analog scales. The EORTC QLQ-STO22 with a 22-item stomach cancer-specific questionnaire was also used. It incorporates five hypothesized scales-(dysphasia, eating restrictions, pain, reflux and anxiety) and four single items (having a dry mouth, body image, taste, and hair loss) covering disease and treatment-related symptoms and specific emotional consequences of gastric cancer.12 All instruments of the questionnaire were administered preoperatively and postoperatively at seven days, 30 days, 90 days and yearly. Those time points were chosen at usual follow-up schedule for every gastrectomized patients in our institute, to maximize compliance for the questionnaire, and to compare other parameters at the same time.
4. Statistical analyses The EORTC QLQ-C30 symptom subscale and the EORTC QLQ-STO22 subscale scores are reported using a scale from 0 to 100. Statistical analyses of the QOL outcomes evaluated the differences between the LADG and the ODG groups with respect to the overall changes from the preoperative scores (baseline) to those obtained at follow-up. To adjust for possible baseline differences, we included the baseline values in the model. All comparisons between groups were based on 'intent-to-treat' analyses in which patients were analyzed according to their assigned treatment group. Categorical variables were compared using the χ2 test, and continuous variables were analyzed using the Student's t-test. Analysis of Covariance (ANCOVA) with repeated measures was used to compare the two groups of patients with respect to overall changes in their short term quality of life after the surgery. The SAS (SAS Institute Inc., Cary, NC, USA) program called 'PROC GLM' was used.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of stomach
* Age: 18-80 years
* Performance status: ECOG 0-1
* Informed consent should be signed
* EGD finding of early gastric cancer
* EUS finding of mucosa and submucosa cancer
* The location of the tumor should be antrum, angle, lower body in greater curvature in UGIS
* No evidence of distant metastasis in abdomen CT, and chest PA
* Regional lymph node metastasis confined to perigastric node (N1) in CT and EUS

Exclusion Criteria:

* Any comorbidity obviating major surgery
* Contraindication of laparoscopy: severe cardiac disease, abdominal wall hernias, diaphragmatic hernias, uncorrected coagulopathies, portal hypertension, pregnancy
* Previous upper abdominal operation
* Indication of EMR: well or moderately differentiated adenocarcinoma, less than 2 cm in EGC type I and IIa, less than 1cm in EGC type IIb and IIc, no ulceration
* Complicated case needed to get emergency operation
* Any accompanying surgical condition needed to be performed in same time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2003-06; Primary Completion 2005-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
5 year disease free survival | 1week, 1 month, 3 months, 6 months,1 year, 2 years, 3 years,4 years, & 5 years
  Laparoscopy assisted distal gastrectomy could be accepted as a oncologically safe and effective treatment if 5 year disease free survival is not inferior compared to open distal gastrectomy. Any recurrence event will be followed up through regular physical and history examinations, imaging by abdominal computed tomography,esophagogastroduodenoscopy and tumor marker like CEA, CA 19-9,and CA 72-4

SECONDARY OUTCOMES:
Quality of life measured by EORTC QLQ | 1week, 1 month, 3 months, 6 months,1 year, 2 years, 3 years,4 years, & 5 years
  EORTC C-30 & Sto-22 engines were measured by self administered questionnaires to compare quality of life between two surgery. Short term evaluation at 3 months, and long term evaluation after 5 years will be done.
Surgical complications | 1 week, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Any surgical complications during and after operation will be compared. Long term complications will be monitored also.
Postoperative surgical outcome | within 1 week daily
  day of starting bowel movement, day of defevescence, hospital stay, white blood cell counts, C reactive protein, amount of transfusion
Overall survival | 1week, 1 month, 3 months, 6 months,1 year, 2 years, 3 years,4 years, & 5 years
  Overall survival regardless of cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, M.D., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Kim YW, Baik YH, Yun YH, Nam BH, Kim DH, Choi IJ, Bae JM. Improved quality of life outcomes after laparoscopy-assisted distal gastrectomy for early gastric cancer: results of a prospective randomized clinical trial. Ann Surg. 2008 Nov;248(5):721-7. doi: 10.1097/SLA.0b013e318185e62e. PMID 18948798
- [Derived] Kim YW, Yoon HM, Yun YH, Nam BH, Eom BW, Baik YH, Lee SE, Lee Y, Kim YA, Park JY, Ryu KW. Long-term outcomes of laparoscopy-assisted distal gastrectomy for early gastric cancer: result of a randomized controlled trial (COACT 0301). Surg Endosc. 2013 Nov;27(11):4267-76. doi: 10.1007/s00464-013-3037-x. Epub 2013 Jun 21. PMID 23793805
- See also: The official web site of National Cancer Center — http://www.ncc.re.kr